CLINICAL TRIAL: NCT01328509
Title: Zinc and Inflammation in Sepsis
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: UK Intensive Care Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11/AL/0137
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Sepsis
Keywords: Zinc
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral whole blood will be sampled from an indwelling arterial line and plasma will be separated. Peripheral blood mononuclear cells will be separated using single density gradient centrifugation and RNA extracted. Nuclear extracts of MNC will also be prepared.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis: Patients with sepsis
- Control: Patients with no clinical evidence of sepsis, but who are critically ill

SUMMARY:
The purpose of the proposed project is to investigate measures of zinc status in relation to oxidative stress and inflammation in patients with sepsis. We hypothesise that zinc depletion can modulate inflammatory responses, leading to increased oxidative stress and mitochondrial dysfunction.

Sepsis is a severe infection is the leading cause of death in critically ill patients [1]. Zinc deficiency impairs overall immune function and resistance to infection [2]. In vitro exposure of monocytes to lipopolysaccharide (LPS) leads to decreased cellular zinc content [3] and zinc redistribution has been shown in human volunteers in response to LPS [4]. Zinc depletion occurs in hospitalized patients including those with infections, the elderly, alcoholics, trauma or burns [5-8], conditions which are common among critically ill patients with sepsis. In a mouse model of sepsis, zinc depletion prior to sepsis resulted in more inflammation and more severe organ injury and increased mortality [9]. In patients with sepsis, early feeding with zinc resulted in faster recovery of organ function compared with control [10]. Zinc status is likely to be compromised in the critically ill and that zinc depletion may affect inflammatory responses and recovery.

Although zinc is not an antioxidant itself, it binds to metallothionein [11] and zinc supplementation decreases oxidative stress [12]. Oxidative stress has been consistently reported in patients with sepsis [13-15]. We have recently shown that protection of mitochondrial function with antioxidants can reduce organ damage in rats [16]. Pentraxin-3 is an inflammatory marker which is regulated in part by antioxidants and plays a key role in innate immunity [17].

The consequences of zinc deficiency may relate, in part, to its effects on nuclear factor NFκB, a transcription factor crucial to the signalling networks involved in sepsis [18]. Higher NFκB activity is associated with increased mortality in patients with sepsis [19,20]. It is likely that compromised antioxidant defences and inflammation occurs as a consequence of zinc deficiency.

We propose to measure plasma zinc and metallothionein mRNA status in relation to inflammatory markers including key cytokines, pentraxin-3, markers of oxidative stress and antioxidant status in patients with sepsis.

DETAILED DESCRIPTION:
Following ethical approval consent will be sought from either the patient, or assent from a near relative. Successive patients admitted to the Intensive Care Unit at Aberdeen Royal Infirmary who fulfil the following criteria for sepsis, given below, within a 24h time window, will be included.

* Clinical suspicion or evidence of acute infection
* SIRS defined by two or more of the following:

  1. Core temperature <36 degrees C or >38 degrees C
  2. Tachycardia; heart rate > 90 beats/min.
  3. Tachypnoea; respiratory rate > 20 breaths/min or mechanical ventilation
  4. White blood count >12 x 109/l or <4 x 109/l

In this pilot study we will recruit 20 patients with sepsis and 20 critically ill patients with no clinical suspicion of sepsis. Patients will be excluded if they are <16 years, pregnant or lactating, HIV positive, receiving corticosteroids or other known immuno-modulatory drugs (including statins), have cancer or autoimmune disorders or if consent/assent is refused.

Blood samples will be obtained on Days 1,2, 5, 10 and 14 of the ICU stay. Peripheral whole blood will be sampled from an indwelling arterial line and plasma will be separated for analysis of plasma zinc using atomic absorption spectroscopy. Plasma interleukin-6 (IL-6) and pentraxin-3 (PTX3) will be measured using enzyme immunoassay and total antioxidant capacity and lipid hydroperoxides will be measured colourimetrically [17]. Peripheral blood mononuclear cells (MNC) will be separated using single density gradient centrifugation, RNA extracted and metallothionein mRNA measured using qPCR [21]. Nuclear extracts of MNC will be prepared and nuclear factor kappa B (NFκB)activation measured using an enzyme immunoassay [17].

ELIGIBILITY:
Patients with sepsis

Inclusion Criteria:

* admitted to ICU with clinical suspicion or evidence of acute infection PLUS two or more of the following:

  1. Core temperature <36 degrees C or >38 degrees C
  2. Tachycardia; heart rate > 90 beats/min.
  3. Tachypnoea; respiratory rate > 20 breaths/min or mechanical ventilation
  4. White blood count >12 x 10 9/l or <4 x 10 9/l

     Control patients
* admitted to ICU with no clinical evidence or suspicion of infection

Exclusion Criteria:

* under 16 years old
* pregnant or lactating
* HIV positive
* receiving corticosteroids or other known immuno-modulatory drugs
* treated with statins in the last month
* have cancer
* have autoimmune disorders
* consent/assent is refused

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Successive patients admitted to the Intensive Care Unit at Aberdeen Royal Infirmary who fulfil the following criteria for sepsis, given below, within a 24h time window.
  • .
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Plasma zinc concentration | 14 days
  Plasma zinc will be measured in patients with sepsis and non-spetic critically ill control patients.

SECONDARY OUTCOMES:
Interleukin-6 | 14 days
  The relationship between IL-6 and plasma zinc
Pentraxin-3 | 14 days
  The relationship between PTX-3 and plasma zinc
Plasma lipid peroxide | 14 days
  The relationship between LPO and plasma zinc
Plasma total antioxidant capacity | 14 days
  The relationship between TAC and plasma zinc
Metallothionein mRNA | 14 days
  Change in MTmRNA in mononuclear leucocytes in relation to plasma zinc and inflammatory markers
Nuclear factor kappa B | 14 days
  Change in NFkB in nuclear extracts from mononuclear cells in relation to plasma zinc

CONTACTS AND LOCATIONS:
Overall Officials: Helen Galley, PhD, Principal Investigator — University of Aberdeen; Nigel Webster, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom

REFERENCES:
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Rink L, Gabriel P. Zinc and the immune system. Proc Nutr Soc. 2000 Nov;59(4):541-52. doi: 10.1017/s0029665100000781. PMID 11115789
- [Background] Goode HF, Rathbone BJ, Kelleher J, Walker BE. Monocyte zinc and in vitro prostaglandin E2 and interleukin-1 beta production by cultured peripheral blood monocytes in patients with Crohn's disease. Dig Dis Sci. 1991 May;36(5):627-33. doi: 10.1007/BF01297030. PMID 2022165
- [Background] Gaetke LM, McClain CJ, Talwalkar RT, Shedlofsky SI. Effects of endotoxin on zinc metabolism in human volunteers. Am J Physiol. 1997 Jun;272(6 Pt 1):E952-6. doi: 10.1152/ajpendo.1997.272.6.E952. PMID 9227437
- [Background] Goode HF, Penn ND, Kelleher J, Walker BE. Evidence of cellular zinc depletion in hospitalized but not in healthy elderly subjects. Age Ageing. 1991 Sep;20(5):345-8. doi: 10.1093/ageing/20.5.345. PMID 1755390
- [Background] Schmuck A, Roussel AM, Arnaud J, Ducros V, Favier A, Franco A. Analyzed dietary intakes, plasma concentrations of zinc, copper, and selenium, and related antioxidant enzyme activities in hospitalized elderly women. J Am Coll Nutr. 1996 Oct;15(5):462-8. doi: 10.1080/07315724.1996.10718625. PMID 8892172
- [Background] Goode HF, Kelleher J, Walker BE. The effects of acute infection on indices of zinc status. Clin Nutr. 1991 Feb;10(1):55-9. doi: 10.1016/0261-5614(91)90082-n. PMID 16839895
- [Background] Berger MM, Cavadini C, Chiolero R, Dirren H. Copper, selenium, and zinc status and balances after major trauma. J Trauma. 1996 Jan;40(1):103-9. doi: 10.1097/00005373-199601000-00019. PMID 8576970
- [Background] Knoell DL, Julian MW, Bao S, Besecker B, Macre JE, Leikauf GD, DiSilvestro RA, Crouser ED. Zinc deficiency increases organ damage and mortality in a murine model of polymicrobial sepsis. Crit Care Med. 2009 Apr;37(4):1380-8. doi: 10.1097/CCM.0b013e31819cefe4. PMID 19242332
- [Background] Beale RJ, Sherry T, Lei K, Campbell-Stephen L, McCook J, Smith J, Venetz W, Alteheld B, Stehle P, Schneider H. Early enteral supplementation with key pharmaconutrients improves Sequential Organ Failure Assessment score in critically ill patients with sepsis: outcome of a randomized, controlled, double-blind trial. Crit Care Med. 2008 Jan;36(1):131-44. doi: 10.1097/01.CCM.0000297954.45251.A9. PMID 18007263
- [Background] Bell SG, Vallee BL. The metallothionein/thionein system: an oxidoreductive metabolic zinc link. Chembiochem. 2009 Jan 5;10(1):55-62. doi: 10.1002/cbic.200800511. PMID 19089881
- [Background] Prasad AS. Clinical, immunological, anti-inflammatory and antioxidant roles of zinc. Exp Gerontol. 2008 May;43(5):370-7. doi: 10.1016/j.exger.2007.10.013. Epub 2007 Nov 1. PMID 18054190
- [Background] Goode HF, Cowley HC, Walker BE, Howdle PD, Webster NR. Decreased antioxidant status and increased lipid peroxidation in patients with septic shock and secondary organ dysfunction. Crit Care Med. 1995 Apr;23(4):646-51. doi: 10.1097/00003246-199504000-00011. PMID 7712754
- [Background] Cowley HC, Bacon PJ, Goode HF, Webster NR, Jones JG, Menon DK. Plasma antioxidant potential in severe sepsis: a comparison of survivors and nonsurvivors. Crit Care Med. 1996 Jul;24(7):1179-83. doi: 10.1097/00003246-199607000-00019. PMID 8674332
- [Background] Galley HF, Howdle PD, Walker BE, Webster NR. The effects of intravenous antioxidants in patients with septic shock. Free Radic Biol Med. 1997;23(5):768-74. doi: 10.1016/s0891-5849(97)00059-2. PMID 9296454
- [Background] Lowes DA, Thottakam BM, Webster NR, Murphy MP, Galley HF. The mitochondria-targeted antioxidant MitoQ protects against organ damage in a lipopolysaccharide-peptidoglycan model of sepsis. Free Radic Biol Med. 2008 Dec 1;45(11):1559-65. doi: 10.1016/j.freeradbiomed.2008.09.003. Epub 2008 Sep 17. PMID 18845241
- [Background] Hill AL, Lowes DA, Webster NR, Sheth CC, Gow NA, Galley HF. Regulation of pentraxin-3 by antioxidants. Br J Anaesth. 2009 Dec;103(6):833-9. doi: 10.1093/bja/aep298. Epub 2009 Oct 28. PMID 19864306
- [Background] Otsu K, Ikeda Y, Fujii J. Accumulation of manganese superoxide dismutase under metal-depleted conditions: proposed role for zinc ions in cellular redox balance. Biochem J. 2004 Jan 1;377(Pt 1):241-8. doi: 10.1042/BJ20030935. PMID 14531733
- [Background] Paterson RL, Galley HF, Dhillon JK, Webster NR. Increased nuclear factor kappa B activation in critically ill patients who die. Crit Care Med. 2000 Apr;28(4):1047-51. doi: 10.1097/00003246-200004000-00022. PMID 10809280
- [Background] Bohrer H, Qiu F, Zimmermann T, Zhang Y, Jllmer T, Mannel D, Bottiger BW, Stern DM, Waldherr R, Saeger HD, Ziegler R, Bierhaus A, Martin E, Nawroth PP. Role of NFkappaB in the mortality of sepsis. J Clin Invest. 1997 Sep 1;100(5):972-85. doi: 10.1172/JCI119648. PMID 9276714
- [Background] Kwon CS, Kountouri AM, Mayer C, Gordon MJ, Kwun IS, Beattie JH. Mononuclear cell metallothionein mRNA levels in human subjects with poor zinc nutrition. Br J Nutr. 2007 Feb;97(2):247-54. doi: 10.1017/S0007114507328614. PMID 17298692
- [Background] Goode HF, Kelleher J, Walker BE. Zinc concentrations in pure populations of peripheral blood neutrophils, lymphocytes and monocytes. Ann Clin Biochem. 1989 Jan;26 ( Pt 1):89-95. doi: 10.1177/000456328902600114. PMID 2735753
- [Derived] Mertens K, Lowes DA, Webster NR, Talib J, Hall L, Davies MJ, Beattie JH, Galley HF. Low zinc and selenium concentrations in sepsis are associated with oxidative damage and inflammation. Br J Anaesth. 2015 Jun;114(6):990-9. doi: 10.1093/bja/aev073. Epub 2015 Mar 31. PMID 25833826